CLINICAL TRIAL: NCT02536222
Title: Accelerating the Reduction of Malaria Transmission in Kanel, Ranérou and Linguère Districts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: National malaria Control Program of Senegal (Unknown); Regional and district health authorities of Matam and Louga regions and Kanel Ranerou and Linguere districts of Senegal (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 762488-1
Record Dates: First submitted 2015-08-05; First posted 2015-08-31 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reactive case investigation : FT/FDA with DHA-PQ (Experimental): All consenting household members eligible to receive DHA-PQ and living in a household where anyone in the household tests positive with a malaria rapid diagnostic test (RDT) will receive the age-appropriate treatment dose of DHA-PQ. If no one in the household tests RDT positive then no one in the household will receive DHA-PQ.
  Interventions: Other: Case investigation of malaria passively detected cases with FT/FDA
- No Intervention: Standard of Care (Control) (No Intervention): The standard of care arm will have the standard of care offered by the Ministry of Health which applies to all arms. This includes available mosquito net coverage and passive case detection of individuals seeking treatment from a health provider at a health post or community.

INTERVENTIONS:
Other: Case investigation of malaria passively detected cases with FT/FDA — Systematic reactive malaria case investigation will be performed in all villages of the six intervention health posts. All malaria cases passively detected in a health post or in the community and confirmed with a positive rapid diagnostic test (RDT) will be considered an index case and will be investigated. A team (field worker and community health worker) will visit the household of the index case and the five closest households (in a 100 meter radius) and will test by RDT all the consenting individuals living in the households. Any households with at least one positive RDT (including the index case) will receive a systematic focal drug administration (FDA) treatment with DHAP through which all members will be treated.
  Arms: Reactive case investigation : FT/FDA with DHA-PQ

SUMMARY:
The work will be conducted in six health posts in the regions of Matam (Kanel and Ranérou districts) and Louga (Linguère district), that were selected in 2014 on the basis of the malaria incidence rate, the heterogeneity of transmission between villages in the health post catchment areas, their proximity, and the availability of historical data from before 2014. Malaria elimination strategies were already implemented in the same health posts in 2014 and are still ongoing, thus this protocol aims to strengthen these activities. Seven health posts with similar characteristics but with a slightly lower incidence rate were chosen as controls. It will be implemented in all villages in the six intervention health posts and it will consist of investigating all passively detected cases (index cases) and conducting focal test and focal drug administration (FT/FDA) with dihydroartemisinin-piperaquine (DHAP) in all index case and neighboring households with a positive RDT. All household members in households with a positive RDT will be treated, regardless of their RDT results. Impact of the enhanced Step D on malaria incidence and prevalence will be evaluated using before-after comparison and compared to the change in the control health posts and the operational aspects will be assessed for subsequent scale up.

DETAILED DESCRIPTION:
1. Introduction:

   During the last decade, 34 countries that have set the objective of freeing themselves from malaria, have obtained remarkable success in reducing the burden of the disease to very low levels that could represent a starting point to elimination programs leading to complete elimination. This remarkable success led several other countries to develop malaria elimination programs supported by the Global Malaria Action Plan of the Roll Back Malaria Partnership: "For a malaria-free world" which has for objective to eliminate malaria in at least 35 endemic countries by 2030. However, the transition from a strategy of malaria control toward a program centered on elimination has not yet been documented. PATH collaborates with the PNLP and regional and district health authorities to produce evidence that allows to make decisions on a model of reduction of malaria transmission in health posts. To that effect, a set of strategies will be put in place and evaluated to efficiently identify and eliminate malaria infections. Thus, zones freed from the disease will be documented. In Senegal, the epidemiological profile of malaria presents the conditions for disease elimination in the North and North-central areas of the country. Since 2012, the National Malaria control program, with support from PATH, has the objective of reducing Plasmodium falciparum transmission in several geographical areas of Saint-Louis, Matam and Louga regions.
2. Goal and Objective:

   The goal of the proposed work is to contribute to the national effort of malaria pre-elimination in Senegal, in line with the National Malaria control program's 2014-2018 strategic framework.

   The main objective is to strengthen the implementation of malaria case investigation in Linguère, Ranérou and Kanel districts, to evaluate operational aspects of scaling up the strategy and to evaluate the impact on malaria transmission to guide evidence-based decision-making.
3. Sites:

   The work will be conducted in six health posts in the regions of Matam (Kanel and Ranérou districts) and Louga (Linguère district), that have been chosen on the basis of the malaria incidence rate, the wide differences of transmission between villages in the health post catchment areas, their proximity and the availability of historical data from before 2014. Malaria elimination strategies were already implemented in the same health posts in 2015, thus this protocol aims to strengthen these activities. Seven health posts with similar characteristics were chosen as controls.
4. Study design A quasi-experimental study design will be used to evaluate the impact of the intervention. The incidence of malaria cases and the prevalence of parasitemia will be compared before and after the intervention and between the intervention and the control areas (difference-in-differences). Cross-sectional surveys will be conducted to estimate the parasitemia prevalence with RDT at the beginning and at the end of the high transmission season in intervention and in control areas.
5. Methodology Systematic malaria case investigation will be performed in all villages of the 6 intervention health posts. All malaria cases passively detected in a health post or in the community and confirmed with a positive rapid diagnostic test (RDT) will be considered an index case and will be investigated. A team (field worker and community health worker (DSDOM)) will visit the household of the index case and the 5 closest households (in a 100 m radius) and will test by RDT all the individuals living in the households. Any households with at least one positive RDT (including the index case) will receive a systematic focal drug administration (FDA) treatment with dihydro-artemisinin-piperaquine (DHA-PQ)
6. Duration:

The study is scheduled to last one year.(July 2015-June 2016).

ELIGIBILITY:
Inclusion Criteria:

* Signs the informed consent form
* Aged more than 2 months
* Resident member of the selected household
* Does not present any severity symptoms

Exclusion Criteria:

* Refuses to sign the informed consent form
* Aged less than 2 months
* Is not a resident member of the selected household
* Presents severity symptoms

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20379 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of passively detected malaria cases | one malaria transmission season (up to 5 months)
  Incidence of passively detected RDT-confirmed malaria cases among individuals older than 2 months (at the health posts or by community health workers), collected through the rapid reporting system already in place. Every week, health facility workers submit basic information on malaria burden, that is entered into DHIS2 (district health information system) at the district level. The quality of the rapid reporting system will be monitored through routine data quality audits (comparing health post registers with submitted data) and continuous monitoring of the data submitted to DHIS2. The estimated enrollment is 30 000 individuals. A comparison before and after the intervention and between interventions and control villages will be done using a difference-in-difference analysis.

SECONDARY OUTCOMES:
Prevalence of Plasmodium falciparum parasitaemia | At the begining (one month after the first rain) and the end (one month after the last rain) of the transmission season
  Prevalence of infection by RDT/polymerase chain reaction (PCR): will be measured during cross-sectional surveys at the beginning and at the end of the transmission season. 16,000 participants are expected to take part in both cross sectional surveys. The prevalence by PCR will only be available later when the laboratory results become available. A comparison before and after the intervention and between interventions and control villages will be done using a difference-in-difference analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- six health posts in Kanel, Linguère and Ranérou districts, Oudallaye, Mbem-Mbem, Salalatou, Doundé, Nianghana, Gassane, Louga and Matam, Senegal